CLINICAL TRIAL: NCT06888492
Title: An Open-label, Dose-escalation Study to Evaluate the Safety and Efficacy of Intravitreal EXG202 Injection in Patients with Wet (neovascular) Age-related Macular Degeneration (wAMD)
Brief Title: To Evaluate the Safety and Preliminary Efficacy of Intravitreal EXG202 Injection in Patients with Wet (neovascular) Age-related Macular Degeneration (wAMD)
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hangzhou Jiayin Biotech Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EXG202-011
Record Dates: First submitted 2025-03-14; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Wet Age-related Macular Degeneration (wAMD); Wet Age-related Macular Degeneration
Keywords: wAMD; AAV

STUDY DESIGN:
Intervention Model Description: Dose escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Dose escalation-Cohort A (Experimental): Dose 1 :Administered via intravitreal injection
  Interventions: Biological: EXG202
- Experimental: Dose escalation-Cohort B (Experimental): Dose 2 :Administered via intravitreal injection
  Interventions: Biological: EXG202

INTERVENTIONS:
Biological: EXG202 — EXG202 is a gene therapy product for the treatment of wet (neovascular) age-related macular degeneration（wAMD） with a single intravitreal injection and administration.

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability and efficacy of intravitreal injection of EXG202 in subjects with neovascular age-related Macular Degeneration (nAMD).

DETAILED DESCRIPTION:
EXG 202 is a gene therapy product developed for the treatment of neovascular age-related macular degeneration (nAMD). Neovascular AMD is the main cause of blindness among elderly individuals. The available therapies for treating nAMD require life-long intravitreal (IVT) injections every 4-12 weeks to maintain efficacy. Administration of EXG202 has the potential to treat nAMD by providing durable expression of therapeutic levels of intraocular protein and maintaining the vision of patients. EXG 202 is designed to reduce the current treatment burden which often results in undertreatment and vision loss in patients with nAMD receiving anti-VEGF therapy in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥50 years old;
2. The study eye must meet the following criteria:

   A. Diagnosed of wAMD and current active lesions; active, defined as the presence of any of the following lesions in the macular area upon OCT examination: a) intraretinal hemorrhage or fluid; b) subretinal fluid; c) subretinal hemorrhage; B. The BCVA score tested during screening using the ETDRS eye chart (see Appendix 3 for details) must be between 73-19 letters (including boundary values), (equivalent to Snellen visual acuity of 20/40 to 20/400);
3. Clinically meaningful response to standard anti-VEGF therapy within 6 months before screening or during the lead-in period of screening.
4. The subject has clear refractive media and sufficient pupil dilation at the time of screening to obtain high-quality retinal images for confirmation of diagnosis;
5. Subjects (including male subjects) have no pregnancy plans during the screening period and the entire trial period and voluntarily take effective contraceptive measures and have no sperm or egg donation plans;
6. Voluntarily participate in this clinical trial, understand the research procedures and sign the informed consent form before screening; have good compliance and are willing to abide by the research procedures.

Exclusion Criteria:

1. The study eye has any eye disease other than wAMD that may affect central vision and/or macular detection (such as macular hole, macular epiretinal membrane, etc.);
2. The study eye has a history of retinal detachment or retinal detachment during the screening period (such as rhegmatogenous retinal detachment, tractional retinal detachment, etc.);
3. The study eye has MNV caused by reasons other than wAMD (such as diabetic retinopathy, pathological myopia, retinal vein occlusion, angioid streak disease, ocular histoplasmosis, trauma, etc.), and a history of macular pathology unrelated to wAMD;
4. The study eye plans to undergo any intraocular surgery during the study period;

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-03-28 (Estimated); Primary Completion 2026-04-25 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability after EXG202 injection | up to 52 weeks after treatment
  Frequency, type, and intensity of ocular and non-ocular Adverse Events (AEs) and serious adverse events (SAE) at Week 52, to explore the maximum tolerated dose (MTD)

SECONDARY OUTCOMES:
To evaluate the efficacy after EXG202 injection | up to 52 weeks after treatment
  the Best Corrected Visual Acuity (BCVA) change from baseline
To evaluate the efficacy after EXG202 injection | 52 weeks following EXG202 treatment.
  The optical coherence tomography (OCT ).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Hebei Eye Hospital, Xingtai, Hebei
  - The Fourth Affiliated Hospital of Zhejiang University School of Medicine, Yiwu, Zhejiang

IPD SHARING:
Plan to Share IPD: No